CLINICAL TRIAL: NCT02979314
Title: Overlapping Cortical Networks of Illusory and Mental Body Transformations
Brief Title: The Influence of GVS on Mental Transformation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-00464
Record Dates: First submitted 2016-08-23; First posted 2016-12-01 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Focus of Study: Higher Cognition and the Vestibular System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Galvanic Vestibular Stimulation (Experimental): A standard placement of the electrodes will be used for GVS and sham, placed on the mastoids. Weak currents up to maximally 3 mA will be used (tested before in each participant individually, and expected mean current will be around 1.5 mA). Previous studies have used Magnetic Resonance (MR) compatible GVS without reporting any discomfort for the participants, however weak sensations of nausea could be possible and in case that they are disturbing for the participants the experiment will be aborted. Continuous stimulation for up to 30min with intensities of 1-1.5 mA is generally considered as safe and free of any considerable side effects.
  Interventions: Device: Galvanic Vestibular Stimulation

INTERVENTIONS:
Device: Galvanic Vestibular Stimulation — The investigators aim to study the influence of Galvanic Vestibular Stimulation on the brain mechanisms underlying illusory self-motion and its influence on egocentric mental transformation. As a control condition sham stimulation will be applied by the same device within the same participants in different trials. Participants should not note the difference.

SUMMARY:
Corroboratory behavioral evidence showed interaction effects between vestibular stimulation and egocentric transformation.

The investigators here examine in healthy participants, whether there are shared brain mechanisms underlying galvanic vestibular stimulation, illusory self-motion and egocentric transformation, as well as their interaction.

It is hypothesized that the GVS induced illusory self-motion dampens the ability to perform egocentric mental transformation.

DETAILED DESCRIPTION:
Theories of embodied mental rotation suggest overlapping processes between real body and egocentric mental transformations. Corroboratory behavioral evidence showed interaction effects between vestibular stimulation and egocentric transformation. Yet, no study so far has investigated which cortical areas are involved in vestibular processing and/or illusory self-motion and mental transformation tasks within the same participants. This however seems crucial, as important individual differences exist for both mental transformation abilities as well as in subjective perception of artificial vestibular stimulation.

The primary objective is to reveal which brain area(s) are involved in the interaction of illusory self-motion (as induced by galvanic vestibular stimulation (GVS)) and egocentric mental transformation, as compared to no illusory self-motion or object-based mental transformation. It is hypothesized that the GVS induced illusory self-motion dampens the ability to perform egocentric mental transformation more than object-based mental transformation.

As previous behavioral studies on such an interaction were always done in a sitting position, a secondary objective is to first replicate previous behavioral mental rotation studies that used GVS, in the Magnetic Resonance (MR) -scanner comparable setting. Moreover, as no brain imaging study so far has investigated subjective illusory motion experience induced by GVS, illusory self-motion will be measured and included in the statistical model to find specific brain regions modulating the illusory self-motion perception.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Written informed consent by the participant
* Right handed

Exclusion Criteria:

* possession of metallic implants, cardiac pacemakers, neuro-stimulators, metal splinter injuries
* claustrophobia
* no ability to lie still in the scanner, e.g. a cold leading to frequent sneezing and subsequent head movements
* history of neurological or psychiatric disorder
* hearing problems
* concomitant medication
* strong motion sensitivity
* vestibular deficits

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen-Level Dependent (BOLD) -signal change in response to egocentric mental transformation | one day
  The Relative BOLD-signal change in response to egocentric mental transformation during GVS versus mental transformation during sham stimulation will be measured in an functional Magnetic Resonance Imaging (fMRI) paradigm

CONTACTS AND LOCATIONS:
Overall Officials: Lars Michels, MD, Principal Investigator — University Hospital Zurich, Div. of Neuroradiology

IPD SHARING:
Plan to Share IPD: Undecided